CLINICAL TRIAL: NCT01157455
Title: Clinical Trial Program of a Medical Instrument Product
Brief Title: A Registry To Evaluate Safety And Effectiveness Of Everolimus Drug Eluting Stent For Coronary Revascularization
Acronym: SEEDS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CCRF Consulting Co., Ltd. (Other)
Responsible Party: Bo Liu, CCRF
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEEDS
Record Dates: First submitted 2010-07-05; First posted 2010-07-07 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-04

CONDITIONS: Coronary Artery Diseases
Keywords: Stent; Coronary artery diseases
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; Clopidogrel; Heparin; bivalirudin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Everolimus Drug Eluting Stent — Implantation
  Other Names: XIENCE(TM) V EECSS; XIENCE(TM) V stent system
Drug: Aspirin — Orally take by 300mg per day at least within 24 hours before index procedure. Orally 100mg indefinitely after the procedure as a part of dual anti-platelet therapy
Drug: Clopidogrel — A loading dose of 300mg must be given at least 6 hours prior to index procedure, or a loading dose of 75mg/d 72 hours prior to index procedure.
  75mg daily for at least 12 months after the procedure as a part of dual anti-platelet therapy.
Drug: Heparin or Bivalirudin — During procedure or in-hospital, Heparin 100u/kg or Bivalirudin may be given,or follow up the standard practice of each site.

SUMMARY:
This is a prospective, multi-center registry to evaluate safety and effectiveness of the Everolimus Drug Eluting Stent for treatment coronary revascularization in Chinese patients with long lesion, small vessel or multi-vessel diseases.

DETAILED DESCRIPTION:
Study Device:The XIENCE V® Everolimus Eluting Coronary Stent System (XIENCE V EECSS or XIENCE V stent system) is a device/drug combination product consisting of either the MULTI-LINK VISION® Coronary Stent System or the MULTI-LINK MINI VISION® Coronary Stent System coated with a formulation containing everolimus, the active ingredient, embedded in a non-erodible polymer. Design:A prospective, multi-center, registry that is designed to enroll Chinese patients with either Long Lesion, or Small Vessel or Multi-Vessel diseases. Purpose:To evaluate the safety and effectiveness of the XIENCE V® everolimus drug eluting stent for coronary revascularization of patients with either long lesion, or small vessel, or multi-vessel diseases. Enrollment:Approximately 1900 patients will be enrolled in at least 45 but up to 51 centers. Mainland China 41 up to 47 centers, Taiwan China 3 centers and Macao China 1 center. This registry is planned to enroll at least 50% of patients with multi-vessel disease. Primary Endpoint:Ischemia-driven Target Vessel Failure (TVF) which is a composite of cardiac death, myocardial infarction (Q and non-Q wave) and target vessel revascularization (TVR) at 12 months post-index procedure. Follow-Up Visits:30 days, 6 months, 12 months, and 24 months post index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥18 of age; male or (non-pregnant and non-breast feeding) female.
2. Diagnosis of stable angina, unstable angina or silent ischemia (evidence of myocardial ischemia).
3. Target lesion is at least length ≥ 25mm (visual estimate); or the number of target lesion is ≥ 2; or target vessel diameter ≤ 2.75mm.
4. At least one target lesion with a diameter stenosis ≥70% (visual estimate)
5. Acceptable candidate for CABG;
6. The patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided written Notice of Informed Consent, appropriate Ethics Committee(EC); and the patient is willing to comply with specified follow-up evaluations.

Exclusion Criteria:

1. Patients have evidence of an Acute Myocardial Infarction within a week prior to the index procedure.
2. Patient has congenital heart disease, severe valve dysfunction, bridge vascular disease, severe heart failure (NYHA ≥ Ⅲ level), or left ventricular ejection fraction ≤ 30%.
3. Patient has undergone previous stenting anywhere within the previous 1 year.
4. Patient has a preoperative renal dysfunction: serum creatinine> 2.0mg/dl (176.82umol / L).
5. Patient has a history of bleeding diathesis or coagulopathy or patients in whom anti-platelet and/or anticoagulant therapy is contraindicated or in which patient will not be able to comply with dual antiplatelet therapy for at least 1 year;
6. Patient has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel/ticlopidine, Prasugrel, stainless steel alloy, cobalt chromium, rapamycin, styrene-butylene-styrene or poly-lactic acid (PLA) polymer, and/or contrast sensitivity that cannot be adequately premedicated; Patient is allergic to contrast agent Sirolimus.
7. Patient has other medical illness (e.g., cancer, known malignancy , congestive heart failure, organ transplant recipient or candidate) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy is less than 12 months.
8. Currently participating in another investigational drug or device study or patient in inclusion in another investigational drug or device study during follow-up
9. Any significant medical condition which in the Investigator's opinion may interfere with the patient's optimal participation in the study; Patient has poor compliance with the judgment of the investigator and can not complete the study as required.
10. Patient who had heart transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1900 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-03 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
TVF | 12 months post-index procedure.
  Ischemia-driven Target Vessel Failure (TVF) which is a composite of cardiac death, myocardial infarction (Q and non-Q wave) and target vessel revascularization (TVR),12 months post-index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Yuejin Yang, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, China

REFERENCES:
- [Derived] Zhang YJ, Zhao YL, Xu B, Han YL, Li B, Liu Q, Su X, Pang S, Lu SZ, Guo XF, Yang YJ. Clinical impact of dual antiplatelet therapy use in patients following everolimus-eluting stent implantation: insights from the SEEDS study. Chin Med J (Engl). 2015 Mar 20;128(6):714-20. doi: 10.4103/0366-6999.152458. PMID 25758261
- [Derived] Xu B, Yang YJ, Han YL, Lu SZ, Li B, Liu Q, Zhu GY, Cui JY, Li L, Zhao YL, Kirtane AJ; SEEDS Investigators. Validation of residual SYNTAX score with second-generation drug-eluting stents: one-year results from the prospective multicentre SEEDS study. EuroIntervention. 2014 May;10(1):65-73. doi: 10.4244/EIJV10I1A12. PMID 24603020